CLINICAL TRIAL: NCT03068897
Title: Ibuprofen Plus Metaxolone, Tizanidine, or Baclofen for Low Back Pain: A Randomized Trial
Brief Title: Ibuprofen Plus Metaxolone, Tizanidine, or Baclofen for Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-7566
Record Dates: First submitted 2017-02-16; First posted 2017-03-03 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — metaxalone; tizanidine; Baclofen; Ibuprofen; Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Medications provided to patients are encapsulated. Medications vials are labelled with investigational stickers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Metaxalone (Active Comparator): Ibuprofen 600mg mg + metaxalone 400-800mg every 8 hours, as needed for low back pain, x 7 days.
  All participants receive a brief educational intervention.
  Interventions: Drug: Metaxalone; Drug: Ibuprofen 600 mg; Behavioral: Educational intervention
- Tizanidine (Active Comparator): Ibuprofen 600mg mg + tizanidine 2-4mg every 8 hours, as needed for low back pain, x 7 days.
  All participants receive a brief educational intervention.
  Interventions: Drug: Tizanidine; Drug: Ibuprofen 600 mg; Behavioral: Educational intervention
- Baclofen (Active Comparator): Ibuprofen 600mg mg + baclofen 10-20 mg every 8 hours, as needed for low back pain, x 7 days.
  All participants receive a brief educational intervention.
  Interventions: Drug: Baclofen; Drug: Ibuprofen 600 mg; Behavioral: Educational intervention
- Placebo (Placebo Comparator): Ibuprofen 600mg mg + placebo, 1 or 2 capsules, every 8 hours, as needed for low back pain, x 7 days.
  All participants receive a brief educational intervention.
  Interventions: Drug: Ibuprofen 600 mg; Behavioral: Educational intervention

INTERVENTIONS:
Drug: Metaxalone — Metaxalone 400-800mg
  Arms: Metaxalone
Drug: Tizanidine — Tizanidine 2-4mg
  Arms: Tizanidine
Drug: Baclofen — Baclofen 10-20mg
  Arms: Baclofen
Drug: Ibuprofen 600 mg — Ibuprofen
Behavioral: Educational intervention — Research personnel will provide each patient with a 15-minute educational intervention. This will be based on NIAMS's Handout on Health: Back Pain information webpage (available at http://www.niams.nih.gov/Health_Info/Back_Pain/default.asp) Research personnel will review each section of the information sheet with the patient and elicit questions.

SUMMARY:
This is a randomized study, based in emergency departments, in which the investigators determine the utility of adding various skeletal muscle relaxants to standard therapy, which consists of ibuprofen and an educational session. Patients will be enrolled at the time of an emergency visit and followed for three months to determine outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Present to ED primary for management of LBP, defined as pain originating between the lower border of the scapulae and the upper gluteal folds. Flank pain, that is pain originating from tissues lateral to the paraspinal muscles, will not be included.
* Musculoskeletal etiology of low back. Patients with non-musculoskeletal etiologies such as urinary tract infection, ovarian cysts, or influenza like illness will be excluded. The primary clinical diagnosis, at the conclusion of the ED visit, must be a diagnosis consistent with non-traumatic, non-radicular, musculoskeletal LBP.
* Patient is to be discharged home. Patients admitted to the hospital are more likely to be treated with parenteral medication and therefore are not appropriate for this study.
* Age 18-64 Enrollment will be limited to adults younger than 65 years because of the increased risk of adverse medication effects in the elderly.
* Non-radicular pain. Patients will be excluded if the pain radiates below the gluteal folds in a radicular pattern.
* Pain duration <2 weeks (336 hours). Patients with more than two weeks of pain are at increased risk of poor pain and functional outcomes.(9)
* Prior to the acute attack of LBP, back pain cannot occur more frequently than once per month. Patients with more frequent back pain are at increased risk of poor pain and functional outcomes.(9)
* Non-traumatic LBP: no substantial and direct trauma to the back within the previous month
* Functionally impairing back pain: A baseline score of > 5 on the Roland-Morris Disability Questionnaire

Exclusion Criteria:

* Not available for follow-up
* Pregnant or breast-feeding
* Chronic pain syndrome defined as use of any analgesic medication on a daily or near-daily basis
* Allergic to or intolerant of investigational medications
* Contra-indications to non-steroidal anti-inflammatory drugs: 1) history of hypersensitivity to NSAIDs or aspirin 2) active or history of peptic ulcer disease, chronic dyspepsia, or active or history of gastrointestinal bleed 3) Severe heart failure (NYHA 2 or worse) 4) hypertension (JNC7 stage 2 or worse) 5) Chronic kidney disease 3 or worse 6) Current use of anti-coagulants 7) Hepatitis 8) Alcoholism
* Contra-indications to muscle relaxants: 1) Concurrent use of centrally acting opioids; 2) Renal impairment; 3) Liver abnormality including cirrhosis or elevated enzymes 4) Use of any of the following medications: fluvoxamine, fluoroquinolones, amiodarone, mexiletine, propafenone, verapamil, cimetidine, famotidine, acyclovir, ticlopidine, oral contraceptive pills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — per patient
Enrollment: 320 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be available

REFERENCES:
- [Derived] Friedman BW, Irizarry E, Solorzano C, Zias E, Pearlman S, Wollowitz A, Jones MP, Shah PD, Gallagher EJ. A Randomized, Placebo-Controlled Trial of Ibuprofen Plus Metaxalone, Tizanidine, or Baclofen for Acute Low Back Pain. Ann Emerg Med. 2019 Oct;74(4):512-520. doi: 10.1016/j.annemergmed.2019.02.017. Epub 2019 Apr 5. PMID 30955985

RESULTS

PARTICIPANT FLOW:
Groups:
- Metaxalone: Ibuprofen 600mg mg + metaxalone 400-800mg every 8 hours, as needed for low back pain, x 7 days.
  All participants receive a brief educational intervention.
  Metaxalone: Metaxalone 400-800mg
  Ibuprofen 600 mg: Ibuprofen
  Educational intervention: Research personnel will provide each patient with a 15-minute educational intervention. This will be based on NIAMS's Handout on Health: Back Pain information webpage (available at http://www.niams.nih.gov/Health_Info/Back_Pain/default.asp) Research personnel will review each section of the information sheet with the patient and elicit questions.
- Tizanidine: Ibuprofen 600mg mg + tizanidine 2-4mg every 8 hours, as needed for low back pain, x 7 days.
  All participants receive a brief educational intervention.
  Tizanidine: Tizanidine 2-4mg
  Ibuprofen 600 mg: Ibuprofen
  Educational intervention: Research personnel will provide each patient with a 15-minute educational intervention. This will be based on NIAMS's Handout on Health: Back Pain information webpage (available at http://www.niams.nih.gov/Health_Info/Back_Pain/default.asp) Research personnel will review each section of the information sheet with the patient and elicit questions.
- Baclofen: Ibuprofen 600mg mg + baclofen 10-20 mg every 8 hours, as needed for low back pain, x 7 days.
  All participants receive a brief educational intervention.
  Baclofen: Baclofen 10-20mg
  Ibuprofen 600 mg: Ibuprofen
  Educational intervention: Research personnel will provide each patient with a 15-minute educational intervention. This will be based on NIAMS's Handout on Health: Back Pain information webpage (available at http://www.niams.nih.gov/Health_Info/Back_Pain/default.asp) Research personnel will review each section of the information sheet with the patient and elicit questions.
- Placebo: Ibuprofen 600mg mg + placebo, 1 or 2 capsules, every 8 hours, as needed for low back pain, x 7 days.
  All participants receive a brief educational intervention.
  Ibuprofen 600 mg: Ibuprofen
  Educational intervention: Research personnel will provide each patient with a 15-minute educational intervention. This will be based on NIAMS's Handout on Health: Back Pain information webpage (available at http://www.niams.nih.gov/Health_Info/Back_Pain/default.asp) Research personnel will review each section of the information sheet with the patient and elicit questions.
Period: Overall Study
Arm/Group | Metaxalone | Tizanidine | Baclofen | Placebo
Started | 80 | 80 | 80 | 80
Completed | 76 | 76 | 79 | 74
Not Completed | 4 | 4 | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metaxalone | Tizanidine | Baclofen | Placebo | Total
Number analyzed (Participants) | 80 | 80 | 80 | 80 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (10) | 40 (11) | 39 (12) | 39 (11) | 39 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 23 | 36 | 133
  Male | 44 | 42 | 57 | 44 | 187
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 80 | 80 | 80 | 80 | 320
Duration of low back pain in hours [Median (Inter-Quartile Range); unit: hours] | 48 [24 to 83] | 48 [24 to 72] | 72 [24 to 114] | 72 [24 to 96] | 60 [24 to 96]

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Impairment as Measured by the Roland Morris Disability Questionnaire (RMDQ)
Description: The Roland Morris Disability Questionnaire (RMDQ) is a 24 item instrument that evaluates the impact of low back pain on one's daily life. It is most sensitive for patients with mild to moderate disability due to acute, sub-acute or chronic low back pain. Each question can be answered as either a "yes" or "no". The score ranges from 0 to 24 where a higher score reflects greater impairment and, therefore, worsening in the quality of life. The change in RMDQ is obtained by subtracting the RMDQ score at one week after discharge from the baseline score.
Time Frame: Baseline and 7 days
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Metaxalone | Tizanidine | Baclofen | Placebo
Number analyzed (Participants) | 76 | 76 | 79 | 74
units on a scale | 10.1 [8.0 to 12.3] | 11.2 [9.2 to 13.2] | 10.6 [8.6 to 12.7] | 11.1 [9.0 to 13.3]

2. Secondary Outcome: Number of Participants Who Experience Change in Low Back Pain
Description: Change is assessed by verbal numerical scale of which 0 represents no pain and 10 represents the worst pain imaginable between the baseline ED visit and the one week follow-up (baseline - 1 week ). The baseline questions will refer to the time period immediately prior to ED presentation (Before you came to the ER today, were you able to…..)
Time Frame: Baseline and 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Metaxalone | Tizanidine | Baclofen | Placebo
Number analyzed (Participants) | 76 | 76 | 79 | 73
Participants | 28 | 25 | 26 | 22

3. Secondary Outcome: Number of Participants With Need for Medication for Low Back Pain
Description: Patients will be asked what medications they have used for low back pain
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Metaxalone | Tizanidine | Baclofen | Placebo
Number analyzed (Participants) | 76 | 76 | 79 | 73
Participants | 49 | 48 | 49 | 46

4. Secondary Outcome: Levels of Disability
Description: Disability will be assessed with the Roland-Morris Disability Questionnaire (RMDQ) where patients are asked to tick a box if they agree with 24 statements regarding their ability to perform certain activities (dressing, housework, walking). If the don't agree with the statement (able to perform those activities) they need to leave the tick-box blank or unchecked. Every agreement (tick) counts as a point and an absolute value is formed (min: 0, max: 24). The higher the value the higher the disability level.
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Metaxalone | Tizanidine | Baclofen | Placebo
Number analyzed (Participants) | 76 | 76 | 79 | 74
units on a scale | 5 [0 to 16] | 3 [0 to 15] | 6 [0 to 16] | 3 [0 to 15]

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Metaxalone | Tizanidine | Baclofen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80 | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 6/80 | 6/80 | 7/80 | 5/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metaxalone (N=80) | Tizanidine (N=80) | Baclofen (N=80) | Placebo (N=80)
Drowsiness (Nervous system disorders) | 2 (2) | 3 (3) | 4 (4) | 2 (2)
Gastrointestinal complaint (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2)
dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
urinary complaint (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT03068897/Prot_SAP_000.pdf